CLINICAL TRIAL: NCT07209228
Title: Investigating the Role of Haptic Feedback in Virtual Reality Learning Environments for Literacy Acquisition
Brief Title: Haptics in Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Anna Queiroz, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20251020
Record Dates: First submitted 2025-09-30; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Literacy; Literacy-language Intervention; Haptics
Keywords: Virtual Reality; Literacy; Haptics; Education
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haptics-integrated Interactive Virtual Reality (Experimental): Participants in this group will receive haptic feedback delivered through haptic gloves with integrated vibration monitors and finger tracking. Each session will last up to 10 minutes, and participants will go through up to 5 sessions
  Interventions: Behavioral: Haptic-Integrated Interactive Virtual Reality Experience
- Control Arm (Active Comparator): Participants in this group will receive the Virtual Reality (VR) delivered through controllers with vibration-based feedback paired with visual and auditory cues, with hand movements. Each session will last up to 10 minutes, and participants will go through up to 5 sessions.
  Interventions: Behavioral: Traditional Virtual Reality Experience (Hand Controllers)

INTERVENTIONS:
Behavioral: Haptic-Integrated Interactive Virtual Reality Experience — Participants will use haptic gloves to interact with the virtual reality experience
  Arms: Haptics-integrated Interactive Virtual Reality
Behavioral: Traditional Virtual Reality Experience (Hand Controllers) — Participants will use traditional hand controllers to interact with the virtual reality experience
  Arms: Control Arm

SUMMARY:
The purpose of this study is to investigate the role of non-invasive wearable haptic feedback, in supporting literacy-focused Virtual Reality (VR) learning environments. The haptic feedback will be delivered through haptic gloves with integrated vibration monitors and finger tracking. The primary objective is to examine how multisensory engagement, specifically the addition of haptic cues, influences learning outcomes such as phonetic recognition, spelling, and reading skills in early learners.

ELIGIBILITY:
Inclusion Criteria:

* Students from elementary to higher education;
* Students aged 6 years old and up.

Exclusion Criteria:

* Students with significant uncorrected vision;
* Students with significant hearing impairments;
* Students with severe cognitive conditions;
* Students with significant neurological conditions;
* Students with significant motor conditions that would prevent safe participation in a VR-based learning activity.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-23 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Literacy Task Performance | Immediately after the intervention session
  Participants' accuracy and completion rates on in-game literacy tasks (e.g., letter recognition, phonetic matching, spelling) recorded during the final session of the intervention. Performance data is automatically logged by the VR platform.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Queiroz, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No